## Official title: Napping, Sleep, Cognitive Decline and Risk of Alzheimer's Disease

NCT#: NCT03256539

**Document date: 09/21/2023** 

## SleepTIGHT Study Protocol

(Sleep Therapeutics Intervention to improve coGnitive HealTh)

Full Study Title: Napping, Sleep, Cognitive Decline and Risk of Alzheimer's Disease

Principal Investigator: Yue Leng, PhD

University of California, San Francisco 675 18th Street San Francisco, CA 94107 Phone: (415) 713-5916

**Sponsor** 

National Institutes of Health

| Title | Napping, Sleep, Cognitive Decline and Risk of Alzheimer's Disease (SleepTIGHT) |
|---|---|
| Study Duration | Trial duration: 9 weeks + follow-up after 24 weeks |
| Study Center | UCSF Psychiatry department |
| Objective | Determine feasibility of online CBT-I in an older adult population (age 65+) |
| Number of Subjects | 40 |
| Diagnosis and Main Inclusion Criteria | <ul> <li>Inclusion Criteria</li> <li>1) Age 65+,</li> <li>2) evidence of MCI, defined as: self-reported quick dementia rating system (QDRS) - derived global clinical dementia rating score of .5,</li> <li>3) adequate visual and auditory acquit to allow neuropsychological texting;</li> <li>4) evidence of subthreshold or clinical insomnia, defined as a score of 8 or more on the insomnia severity index,</li> <li>5) ability to speak understand and write in English, 6) study partner willing to participate,</li> <li>7) capacity to give written informed consent; and</li> <li>8) owns one or more smartphone or tablet devices that can be used to access the internet and to participate in video conferences.</li> </ul> |
| | <ul> <li>1) Self-reported diagnosis by a physician of any major neurologic disease such as Alzheimer's disease, other dementia, Parkinson's disease, multiple sclerosis, epilepsy, Huntington's disease;</li> <li>2) History of brain tumor or significant head trauma (loss of consciousness &gt;30 minutes);</li> <li>3) Evidence (CT or MRI scans within 12 months prior to screening) of brain infarction or other focal lesions; 4) Any comorbid psychiatric conditions or severe personality disorder within the past 2 years (by DSM-V), such as major depression, bipolar disorder, schizophrenia, and other psychotic features;</li> <li>5) Any uncontrolled medical conditions or systemic illness that might lead to difficulty complying with the study protocol;</li> <li>6) Any concomitant treatment that might confound the results (participants must be off all psychotropic medications, including hypnotic medications, and non-pharmacological treatments, for at least 30 days prior to screening);</li> <li>7) History of alcohol or substance abuse within the past 2 years;</li> <li>8) Shift workers; and</li> <li>9) Any inadequately treated primary or secondary sleep disorders</li> </ul> |

#### STUDY PERSONNEL AND ROLES

| Yue Leng, PhD | Principal Investigator | Responsible for all study-related issues |
|---|---|---|
|---|---|---|

#### **Purpose**

In order to address the hypothesis that CBT-I is feasible in patients with MCI, and could potentially improve their sleep quality, slow down cognitive decline, and improve quality of life of patients and caregivers, we will use a parallel-designed randomized controlled trial to pilot test the feasibility and effects of a digital CBT-I treatment program in those with MCI.

This study focuses on testing the validity of this CBT-I program while exploring its preliminary effects on sleep/cognition.

#### **Duration of the Study**

Screening + Intervention + post-study screening: 10 – 13 weeks

Post-treatment follow-up: After 24 weeks

#### Setting

The trial will take place remotely, with all activities and assessments done over phone or Zoom video call or app on smart device.

#### **Description of the Intervention**

We will randomize patients, using computer-generated random numbers, to one of two treatment arms:

a) an FDA-authorized prescription digital CBT-I therapeutic treatment

or

b) an interactive, attention-matched, internet-based placebo control program.

At the beginning of the intervention, study staff will give instructions on the use of the programs via zoom.

Throughout the intervention, study staff will call the participants weekly to give further clarifications and answer questions. Somryst is a 9-week program that delivers digital CBT-I therapeutic content, and can be used on a mobile device, such as a smartphone or tablet. CBT-I is a neurobehavioral treatment which focuses on addressing the maladaptive behaviors, routines, and dysfunctional thoughts that perpetuate sleep problems, regardless of the cause of sleep problems. CBT-I can be conceptualized as six sessions or cores that deliver proven behavioral and cognitive treatment strategies.

#### **Potential Benefits and Risks to Participants**

There will be no direct benefit to the participants from taking part in this study. Taking part in this study may or may not make their health better. While doctors hope that cognitive training therapies will be beneficial, these trainings are still being studied.

Some of the most likely risks of participation in this study include:

- Risk of fatigue/distress: Finding study activities difficult, tiring, time-consuming, anxiety-provoking, frustrating, or boring. Participants are free to decline to answer any questions or to stop at any time. To reduce fatigue, breaks are scheduled during testing and training sessions. Additional breaks will be provided at the participant's request. If the participant appears to be under undue strain, the session will be discontinued.
- Risk of loss of privacy: Participation in research may involve a loss of privacy. Because training takes place in a small group setting, other research subjects within the group may become aware of information that participants would prefer to not be shared outside of the group. Researchers will ask all subjects to keep private all information learned about other group members and to not talk about this information outside of group sessions. However, absolute confidentiality cannot be guaranteed. The researchers will keep information about participants as confidential as possible, but complete confidentiality cannot be guaranteed. On rare occasions, a court has subpoenaed research records. Other University of California personnel may also review or receive information about the participants. Study PI and research staff will retain the participant's research records indefinitely for research purposes. Personal identifiable information (PII) and protected health information (PHI) cannot be used for additional research without additional approval from either the participant or a review committee.
- Unknown risks: The experimental treatments may have risks or side effects that no one knows about yet.
   Members of the research team will inform participants about any new information that may impact their decision to remain in the study.

#### **Recruitment Methods**

Participants are recruited from MyChart patient records, screen in Computerized Patient Record System (CPRS), that meet inclusion criteria. Also, to be used: Research Match and social media recruitment via advertisement on relevant pages associated to CPBH, i.e., Memory and Aging Center.

Keywords checked in medical records:

- Mild Cognitive Impairment
- Age 65 or older
- History of Insomnia
- (Add final ICD-10 terms)

#### Reasons for Participant Withdrawal or Termination

Participants can decide to stop at any time. The study doctor may stop participants from taking part in this study at any time if the doctor believes it is in the participant's best interest, if the participant does not follow study rules, or if the study is stopped

#### **Study Schedule & Procedure Summary**

SCHEDULE OF EVALUATIONS

| ASSESSMENT | Recruitment Pre-screening & Consent | Screening/<br>Assessment | Baseline Measures/<br>Start of Trial | 9 Weeks/<br>End of Trial<br>Follow-up |
|---|---|---|---|---|
| Inclusion/Exclusion | X | | | |
| Criteria | | | | |
| Medical History | X | X | | |
| Insomnia Severity Index | X | Х | | X |
| Pittsburg Sleep Quality | | Х | | Х |
| Index | | | | |
| SF-36 | | | Х | X |
| Epworth Sleepiness Scale | | | Х | Х |
| Quality of Life | | | Х | Х |
| Cognitive function | | | X | X |
| Geriatric Depression Scale | | | Х | |
| 24-h Actigraphy | | | Х | Х |
| (3 days) | | | | |
| Cognitive Assessment | | | Х | X |
| Battery | | | | |

#### **INITIAL CONTACT AND SCREENING**

- 1. Participants, after being identified or reaching out to research team with interest, will be called with initial **contact phone script**, given introductory information about the study, asked to confirm their interest and given the option to fill **consent form** on same call or to schedule follow-up call for consent. IF participant it still interested, consent form is signed, then **ISI questionnaire** is given.
- 2. Followed by appointment for:
  - Baseline Cognitive Assessment Interview: 1 hour via Zoom.
  - Administer the following questionnaires:
    - Pittsburg Sleep quality index
    - Epworth Sleepiness Scale
    - 36-item short-form survey

#### If continued interest, eligible, and consented

- Schedule meeting for briefing via Zoom on Somryst program or placebo condition materials
- Intervention **or** attention-matched placebo program (6 weeks) + Weekly meetings with research team for clarification or assistance with materials and content

#### A. INTERVENTION

Over six weeks, the research team will have scheduled meetings with participants to deliver content and instructions for use of the Somryst

The Somryst program is intended to deliver 6 treatment Cores, with the following specific CBT-I therapy content:

- 1. **Get Ready**: This Core sets the stage for the therapeutic experience. It lets the participant know what they will need to learn and do to improve sleep and sets goals for success.
- 2. **Sleep Window**: This Core focuses on the concept of sleep restriction and identifies a Sleep Window
- a recommended Bedtime and Arising Time the participant should follow.
- 3. **Behaviors**: This Core focuses on stimulus control and establishes guidelines for participants to follow while implementing their Sleep Window.
- 4. **Thoughts**: This Core explains how a participant's thinking can contribute to insomnia. The participant will learn to identify, and shift thought patterns.
- 5. **Education**: This Core helps the participant identify changes to be made in their lifestyle and environment that can promote better sleep.
- 6. **Looking Ahead**: This Core pulls together what the participant has learned, prepares the participant for the future, and teaches them what to do if they experience a relapse. Somryst also includes a daily Sleep Diary in which the participant records information about their sleep.

#### **B. FOLLOW-UP MEASURES**

Once intervention is completed,

- Feedback at the end of trial via survey and phone follow-up (if needed)
- Follow-up (3-day actigraphy & questionnaires + Cognitive Assessments)
- Follow-up at 24 weeks:
- Final follow-up actigraphy watch measurement
- Follow-up of cognitive assessment + questionnaires

#### **OUTCOME MEASURES**

**Primary Outcomes** 

#### **Feasibility**

Proportion of eligible participants consented

- Proportion of participants randomized after baseline assessment
- Number of CBT-I sessions completed
- Adherence/compliance rates
- Follow-up rates
- Missing data (data completeness)
- Time needed to collect and analyze data

#### Acceptability

General study satisfaction Acceptability of intervention Barriers & Burden Qualitative interview

#### **Data Collection and Storage**

Patient information is collected and stored in REDCap.

Once assessments are completed, they will be scored and recorded for later analysis.

#### **Study Outline Graphic**



Figure 1 Outline of study visits and related measurements

#### APPENDIX A.

## SLEEPTIGHT INITIAL CONTACT TELEPHONE SCREENER Full study title - Napping, Sleep, Cognitive Decline and Risk of Alzheimer's Disease

| For those who were pre-screened} |
|---|
| Hello, my name is and I am calling about a research study called SleepTIGHT being conducted at UCSF by Principal Investigator Yue Leng, PhD. |
| Is this a good time? Do you have time to talk for about five to seven minutes to learn briefly about our research study? |
| f no: what would be a good time to call you? (Specify follow-up) |
| If yes: Great! Broadly speaking, this research study is about digital therapeutics to treat sleep problems and improve cognition (Go to BRIEF STUDY OVERVIEW). |
| [For calling back individuals who asked for more information] |
| Hello, my name is Thanks for expressing interest in our research study about sleep, insomnia, and cognitive decline. We appreciate you calling to learn more. The study is being conducted by researchers at the Department of Psychiatry and Behavioral Sciences at UCSF. We wanted to call today to tell you more about the study. Is this a good time? Do you have time to talk for about five to seven minutes to learn briefly about the study? |

#### **BRIEF STUDY OVERVIEW**

Next, I'm going to give you a description of the study. Please stop me if you have any questions.

As mentioned earlier, SleepTIGHT is a study using a digital therapeutic treatment for improving sleep patterns in people with mild impairment in mental processing. This study is unique in that it requires no in-person visits, and the therapy is FDA-approved.

Participants will meet with researchers via phone and videoconference and undergo 6 weeks of (approx. 1 hour) sessions. You will be keeping a sleep diary to track progress and describe sleeping patterns over the course of the study. You will also complete questionnaires that ask about your experience in the program, your quality of life, sleeping habits and mental processing.

The primary goals with treatment are to improve sleep habits which may benefit your mental processing and slow or prevent risk for cognitive decline.

If you are interested in enrolling, you will take part in a few questionnaires and cognitive tests. These are necessary to make sure you are eligible to participate. The screening questions will ask about your quality of life, overall health, mood, and sleep. We also will ask about cognitive function. These questionnaires will take about 45 min - 1 hr. for you to complete.

After this, if you are interested and potentially eligible based on the screening, we will schedule a second appointment via videoconferencing to confirm your eligibility and complete necessary paperwork to begin the study.

Are you still interested in participating? Do you have any questions?

Would you like to do an initial screening for the study, or should I call back later? (it should take an additional 10-15 minutes)

\*\*\*Please note that you are free not to answer any questions you are uncomfortable with, and otherwise please answer as accurately as possible (to best determine your eligibility).

#### SleepTIGHT phone screening script

#### **INTERVIEWER INSTRUCTIONS**

| Read <b>bolded</b> text verbatim. | Answer any questions a | as needed. Record all contacts in the contact log. |
|---|---|---|
| | | unfortunately you are not eligible to participate in this iate and indicate reason for ineligibility]. |
| ☐ Psychiatric condition | edical condition Moderate/severe | ☐ Vision/hearing impairment |
| INTRODUCTION Hi, this is from t | he SleepTIGHT study. | |
| | cted us about the Sleep | <b>Der</b> . E.g., is a UCSF patient who expressed interest in our DTIGHT study. Clarify that the program may also be known as ecessary. |
| Is this a good time for me to should take about 20 minut | _ | tion about your eligibility for the SleepTIGHT study? It |
| □ Yes □ No | | |
| If NO or NOT AVAILABLE: Schedule call-back Date Time: | | |
| If YES:<br>*START HERE IF CONTINUIN | IG CALL* | |
| BACKGROUND INFORMATIO | <u>N</u> | |
| Great! Before we get starte | d, can you please tell n | me your name? [or confirm name if already known] |
| How did you learn about th ☐ UCSF email/letter (1) ☐ F Other (99) | • | (2) $\square$ Physician Referral (3) $\square$ Recruitment Partners (4) $\square$ |

| DEMOGRAPHIC INFORMATION |
|---|
| How old are you? years (enter as current age in whole years; if under 65) |
| Do you identify as male or female? ☐ Male (0) ☐ Female (1) ☐ Other (8) Prefer not to answer (9) |
| Do you identify as Hispanic or Latino? ☐ Hispanic/Latino (1) ☐ Not Hispanic/Latino (0) ☐ Other (7) Prefer not to answer (8) Unknown/Not Reported (9) |
| What race or races do you consider yourself? (check all that apply) ☐ White (1) ☐ Asian (2) ☐ Black or African American (3) ☐ Native Hawaiian or Pacific Islander (4) ☐ American Indian or Alaska Native (5) ☐ Other (8) ☐ ☐ Unknown or Not Reported (9) |
| How many years of school did you complete? Elementary: □ 1 □ 2 □ 3 □ 4 □ 5 □ 6 □ 7 □ 8 High school: □ 9 □ 10 □ 11 □ 12 □ GED College: □ 13 □ 14 □ 15 □ 16 Post-graduate: □ 17 □ 18 □ 19 □ ≥20 □ Not sure |
| ELIGIBILITY CRITERIA |
| Are you able to speak and understand English? □Yes (1) □ No (0) If NO |
| ** Do you have a diagnosis related to memory loss? ☐ Alzheimer's disease (1) ☐ Vascular dementia (2) ☐ Dementia unspecified (3) ☐ Mixed dementia (4) ☐ Mild cognitive impairment (5) ☐ Not sure, but could ask doctor (6) ☐ Other (7) |
| Do you have history of brain tumor or significant head trauma (including for instance, loss of consciousness >30 minutes?) \[ \text{Yes (1)} \text{No (0)} \\ \text{If YES \text{STOP}} \] |
| Has a doctor ever diagnosed you with brain infarction? ☐ Yes (1) ☐ No (0) If YES TOP |

| Has a doctor ever diagnosed you with any severe psychiatric disorders in the past 2 years such as depression, bipolar disorder, schizophrenia or any others? |
|---|
| □Yes (1) □ No (0) |
| If YES STOP |
| IT YES |
| Specify which: |
| Has a doctor ever diagnosed you with any major neurological disease such as Parkinsons' multiple schlerosis, |
| epilepsy, or Huntington's disease? |
| □Yes (1) □ No (0) |
| If YES STOP |
| Specify which: |
| Has a doctor ever diagnosed you with Cognitive Impairment? |
| □Yes (1) □ No (0) |
| Has a doctor ever diagnosed you with Insomnia? |
| □Yes (1) □ No (0) |
| Have you been diagnosed with any sleep disorders (such as sleep apnea, sleep related movement disorders etc.) (yes or no) if yes (have they been treated?) |
| □ No (0) □ Yes (1) If Yes, please describe: If YES |
| Are you currently taking any medications for memory loss or dementia? |
| □Yes (1) □ No (0) |
| *If yes, please indicate which one(s) (check all that apply): |
| ☐ donepezil (Aricept) ☐ galantamine (Razadyne) ☐ rivastigmine (Exelon) |
| ☐ memantine (Namenda) ☐ other |
| Have you been on a steady dose for the past 3 months? |
| □Yes (1) □ No (0) If NO III |
| Are any changes to these medications planned in the next 6 months? |
| $\square$ Yes (1) $\square$ No (0) If NO $\square$ |
| Lifes (1) Lino (0) If NO |
| Have you been on any psychotropic or hypnotic medications within the past 30 days? |
| □ No (0) □ Yes (1) If YES •••• |
| please describe: |
| Do you have a history of alcohol or substance abuse within the past 2 years? |
| □ No (0) □ Yes (1) If YES •••• |

| Are you emplo | yed as a shi | ift-worker? | | | |
|---|---|---|---|---|---|
| □ No (0) | ☐ Yes (1) If | YES | | | |
| Do have vision | or hearing | impairment that co | uld affect your ability to | participate? | |
| □ No (0) | ☐ Yes (1) | If Yes, please des | cribe: | | |
| The next ques | tions will as | k about what device | es you could use for the | online material and ass | essments. |
| - | er mobile de | | amera that can connect<br>ey do not have a mobile | | • |
| ` ' | ` , | , 0 | re information and cont | | |
| • • | | · · | camera access is only n<br>ly a smartphone is neede | | or cognitive |
| Are you willing<br>weeks? | g to participa | ate in the SleepTIGI | IT material for about 35 | minutes on a weekly b | asis over six |
| □ Yes (1) | □ No (0) <sup>1</sup> | | | | |
| - | | ating in another reso | • | | |
| you are eligibl | e for the pai | • | oceed – though we will<br>udy. The next step is to o | | |
| Subject's Initia | ls | ID# | Date | Time | AM/PM |

Please answer the following questions as accurately as possible.

#### PITTSBURGH SLEEP QUALITY INDEX

| INST | ГОІ | $I \cap T$ | | ıc. |
|------|-----|------------|-----|-------------|
| IIVO | IRL | JULI | IUI | <b>45</b> : |

The following questions relate to your usual sleep habits during the past month <u>only</u>. Your answersshould indicate the most accurate reply for the <u>majority</u> of days and nights in the past month. Please answer all questions.

| 1. | During the past mo | onth, what time have yo | ou usually gone to be | d at night? |
|---|---|---|---|---|
| | | BED TIME | · | |
| 2. | During the past mo | onth, how long (in minut | tes) has it usually tak | en you to fall asleep each night |
| | | NUMBER OF N | MINUTES | |
| 3. | During the past mo | onth, what time have yo | ou usually gotten up i | n the morning? |
| | | GETTING UP TI | ME | |
| 4. | | onth, how many hours<br>f hours you spent in be | | you get at night? (This may bedifferent |
| | | HOURS OF S | LEEP PER NIGHT | |
| For eac | h of the remaining q | questions, check the c | one best response. | Please answer <u>all</u> questions. |
| 5. | During the past mo | onth, how often have yo | ou had trouble sleepi | ng because you |
| a) | Cannot get to sleep | p within 30 minutes | | |
| | Not during the last month | Less than<br>once a week | Once or twice<br>_ a week | Three or more times a week |
| b) | Wake up in the mi | ddle of the night or ear | ly morning | |
| | | Less than<br>once a week | Once or twice<br>a week | Three or more times a week |
| c) | Have to get up to | use the bathroom | | |
| | Not during the last month | Less than once a week | Once or twice<br>a week | Three or more times a week |

| d) | ) Cannot breathe comfortably | | | | |
|---|---|---|---|---|---|
| | Not during the last month | Less than once a week | Once or twice a week | Three or more times a week | - |
| e) | Cough or snore loud | dly | | | |
| | Not during the last month | Less than once a week | Once or twice a week | Three or more times a week | - |
| f) | Feel too hot | Less than | Three<br>or | month<br>week | |
| | Not during the | Once or twice | more<br>last | week | annoo a |
| g) | Had bad dreams | Less than | Three<br>or | month<br>week | |
| | Not during the | Once or twice | more<br>last | week | |
| h) | Have pain | Less than | Three<br>or | once<br>a week | a week<br>times a |
| | Not during the | Once or twice | more<br>last<br>month | week | |
| i) | Other reason(s), ple | ease describe | | | |
| Н | ow often during the p | oast month have you ha | d trouble sleeping | because of this? | |
| Not during the Less than Once or twice Three or more last month once a week a week times a week | | | | | |

| 6. | During the past mor | nth, how would you rat | te your sleep quality | overall? | |
|---|---|---|---|---|---|
| | | Very good | | | |
| | | Fairly good | <u> </u> | | |
| | | Fairly bad | _ | | |
| | | Very bad | <del></del> | | |
| 7. | During the past mo the counter")? | nth, how often have y | ou taken medicine t | o help you sleep (prescr | ibed or"over |
| | Not during the last month | Less than once a week | Once or twice<br>a week | Three or more times a week | |
| 8. | During the past mo or engaging in social | | you had trouble stay | ring awake while driving, | eatingmeals |
| | | Less than once a week | | Three or more times a week | |
| 9. | During the past mo | | a problem has it be | en for you to keep up | enough |
| | _ | - | | | |
| | · | olem at all | | | |
| | Only a | very slight problem | | | |
| | Somew | hat of a problem | | | |
| | A very l | big problem | | | |
| 10. | Do you have a bed | partner or roommate? | , | | |
| | No bed | partner or roommate | | | |
| | Partner | r/roommate in other ro | om | | |
| | Partner | in same room, but no | ot in same bed | | |
| | Partner | in same bed | | | |

| a) | Loud snoring | | | |
|---|---|---|---|---|
| | <u> </u> | Less than once a week | | |
| b) | Long pauses betwe | en breaths while asleep | | |
| | Not during the Past month | | | Three or more times a week |
| c) | Legs twitching or je | rking while you sleep | | |
| | | Less than once a week | | Three or more times a week |
| d) | Episodes of disorier | ntation or confusion duri | ng sleep | |
| | | Less than once a week | | Three or more times a week |
| e) | Other restlessness | while you sleep; please | describe | |
| | • | Less than once a week | | Three or more times a week |

If you have a roommate or bed partner, ask him/her how often in the past month you have had . .

#### **Insomnia Severity Index**

The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score. When you have your total score, look at the 'Guidelines for Scoring/Interpretation' below to see where your sleep difficulty fits.

For each question, please CIRCLE the (SAY WHICH choice) number that best describes your answer.

Please rate the CURRENT (i.e., LAST 2 WEEKS) SEVERITY of your insomnia problem(s).

| Insomnia Problem | None | Mild | Moderate | Severe | Very<br>Severe |
|---|---|---|---|---|---|
| Difficulty Falling Asleep | 0 | 1 | 2 | 3 | 4 |
| 2. Difficulty Staying Asleep | 0 | 1 | 2 | 3 | 4 |
| 3. Problems Waking up too early | 0 | 1 | 2 | 3 | 4 |

4. How SATISFIED/DISSATISFIED are you with your CURRENT sleep pattern?

Very Satisfied Satisfied Moderately Satisfied Dissatisfied Very Dissatisfied 0 1 2 3 4

5. How NOTICEABLE to others do you think your sleep problem is in terms of impairing the quality of your life?

Not at all Noticeable A Little Somewhat Much Very Much Noticeable 0 1 2 3 4

| 6. How WORRIED/DISTRESSED are | you about yo | our current sleep | problem? |
|---|---|---|---|
|---|---|---|---|

Not at all Worried A Little Somewhat Much Very Much Worried 0 1 2 3 4

7. To what extent do you consider your sleep problem to INTERFERE with your daily functioning (e.g. daytime fatigue, mood, ability to function at work/daily chores, concentration, memory, etc.) CURRENTLY?

Not at all Interfering A Little Somewhat Much Very Much Interfering 0 1 2 3 4

#### **Guidelines for Scoring/Interpretation:**

Add the scores for all seven items (questions 1 + 2 + 3 + 4 + 5 + 6 + 7) = \_\_\_\_\_\_ your total score

Total score categories:

0–7 = No clinically significant insomnia

8–14 = Subthreshold insomnia

15–21 = Clinical insomnia (moderate severity) 22–28 = Clinical insomnia (severe)

| Note: the Informed Consent does not have to be read word-for-word over the telephone but major points need to be reviewed, including: |
|---|
| Subject Bill of Rights |
| Background and Purpose |
| Study Procedures/Plan |
| Responsibilities |
| Potential Benefits |
| Confidentiality |
| Participation is Voluntary |
| Medical Treatment and Compensation |
| Significant New Information |
| Time Requirements |
| Possible Risks and Discomforts |
| Alternatives to Participate |
| Costs and payments |
| Right of Investigator to Withdraw Subjects |
| Persons to Contact if Questions: |
| Contact Information: Dr. Yue Leng at 415-340-2708 |
| For questions about your rights as a research participant, you can call the UCSF Institutional Review Board at 415-476-1814. |
| Would you be interested in being screened to see if you're eligible for this research? It will take about 30 minutes to go over |
| these questions. |
| It's fine if you want to get back to us later about scheduling a telephone screening appointment [If potential subject |
| wants to schedule phone appointment. When would be a good day and time? |

**Informed Consent Review** [either continuation of above telephone conversation or in later call]

## **Epworth Sleepiness Scale**

Name:\_\_\_\_\_\_Today's date: \_\_\_\_\_

| Your age (Yrs): | Your sex (Ma | ale = M, Female = F): |
|---|---|---|
| How likely are you to doze off or fall | asleep in the following situations, ir | n contrast to feeling just tired? |
| This refers to your usual way of life i | n recent times. | |
| Even if you haven't done some of the | ese things recently try to work out ho | w they would have affectedyou. |
| Use the following scale to choose the | most appropriate number for each | n situation: |
| | 0 = would never doze<br>1 = slight chance of dozing<br>2 = moderate chance of dozing<br>3 = high chance of dozing | |
| It is imp | oortant that you answer each question | on as best you can. |
| Situation | | Chance of Dozing (0-3) |
| Sitting and reading | | |
| Watching TV | | |
| Sitting, inactive in a public place (e.g | a theatre or a meeting) | _ _ |
| As a passenger in a car for an hour w | ithout a break | - _ |
| Lying down to rest in the afternoon w | hen circumstances permit | _ _ |
| Sitting and talking to someone | | _ _ |
| Sitting quietly after a lunch without a | ilcohol | _ _ |
| In a car, while stopped for a few minu | utes in the traffic | _ |

THANK YOU FOR YOUR COOPERATION

© M.W. Johns 1990-97

#### Medical Outcomes Study Questionnaire Short Form 36 Health Survey

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey! For each of the following questions, please (say which choice) eircle the number that best describes your answer.

| 1. In general, would you say your health | |
|------------------------------------------|---|
| is: | |
| Excellent | 1 |
| Very good | 2 |
| Good | 3 |
| Fair | 4 |
| Poor | 5 |
| 2. Compared to one year ago, | |
| Much better now than one year ago | 1 |
| Somewhat better now than one year ago | 2 |
| About the same | 3 |
| Somewhat worse now than one year ago | 4 |
| Much worse now than one year ago | 5 |

3. The following items are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much? (Circle One Number on Each Line)

| | Yes,<br>Limited<br>a<br>Lot (1) | Yes,<br>Limiteda<br>Little<br>(2) | No, Not<br>limited<br>at<br>All (3) |
|---|---|---|---|
| a. <b>Vigorous activities</b> , such as running, lifting heavy objects, participating in strenuous sports | 1 | 2 | 3 |
| b. <b>Moderate activities</b> , such as moving a table, pushing a vacuum cleaner, bowling, or playinggolf | 1 | 2 | 3 |
| c. Lifting or carrying groceries | 1 | 2 | 3 |
| d. Climbing <b>several</b> flights of stairs | 1 | 2 | 3 |
| e. Climbing <b>one</b> flight of stairs | 1 | 2 | 3 |

| f. Bending, kneeling, or stooping | 1 | 2 | 3 |
|------------------------------------|---|---|---|
| g. Walking <b>more than a mile</b> | 1 | 2 | 3 |
| h. Walking <b>several blocks</b> | 1 | 2 | 3 |
| i. Walking <b>one block</b> | 1 | 2 | 3 |
| j. Bathing or dressing yourself | 1 | 2 | 3 |

4. During the **past 4 weeks**, have you had any of the following problems with your work or other regular daily activities **as a result of your physical health**? (Circle One Number on Each Line)

| | Yes | No |
|---|---|---|
| | (1) | (2) |
| a. Cut down the amount of time you spent on work or other activities | 1 | 2 |
| b. <b>Accomplished less</b> than you would like | 1 | 2 |
| c. Were limited in the <b>kind</b> of work or other activities | 1 | 2 |
| d. Had <b>difficulty</b> performing the work or other activities (for example, it took extra effort) | 1 | 2 |

5. During the **past 4 weeks**, have you had any of the following problems with your work or other regular daily activities **as a result of any emotional problems** (such as feeling depressed or anxious)?

### (Circle One Number on Each Line)

| | Yes | No |
|---|---|---|
| a. Cut down the amount of time you spent on work or other | 1 | 2 |
| activities | | |
| b. <b>Accomplished less</b> than you would like | 1 | 2 |
| c. Didn't do work or other activities as <b>carefully</b> as usual | 1 | 2 |

| 6. During the past 4 weeks, to what extent has your physical | |
|---------------------------------------------------------------|---|
| health or emotional problems interfered with your normal | |
| social activities with family, friends, neighbors, or groups? | |
| Not at all | 1 |
| Slightly | 2 |
| Moderately | 3 |
| Quite a bit | 4 |
| Extremely | 5 |

| 7. How much bodily pain have you had during the past 4 | |
|--------------------------------------------------------------|---|
| weeks? | |
| None | 1 |
| Very mild | 2 |
| Mild | 3 |
| Moderate | 4 |
| Severe | 5 |
| Very severe | 6 |
| 8. During the past 4 weeks, how much did pain interfere with | |
| your normal work (including both work outside the home and | |
| housework)? | |
| Not at all | 1 |
| A little bit | 2 |
| Moderately | 3 |
| Quite a bit | 4 |
| Extremely | 5 |

These questions are about how you feel and how things have been with you during the past 4 weeks. For each question, please give the one answer that comes closest to the way you have been feeling. (Circle One Number on Each Line)

9. How much of the time during the **past 4 weeks** . . .

| | All of<br>the<br>Time | Most<br>of the<br>Time | A<br>Good<br>Bit of<br>the<br>Time | Some<br>of the<br>Time | A<br>Little<br>of the<br>Time | None<br>of the<br>Time |
|---|---|---|---|---|---|---|
| a. Did you feel full of pep? | 1 | 2 | 3 | 4 | 5 | 6 |
| b. Have you been a very nervous person? | 1 | 2 | 3 | 4 | 5 | 6 |
| c. Have you felt so down in the dumps that nothing could cheer you up? | 1 | 2 | 3 | 4 | 5 | 6 |
| d. Have you felt calm and peaceful? | 1 | 2 | 3 | 4 | 5 | 6 |
| e. Did you have a lot of energy? | 1 | 2 | 3 | 4 | 5 | 6 |

| | All of<br>the<br>Time | Most<br>of the<br>Time | A<br>Good<br>Bit of<br>the<br>Time | Some<br>of the<br>Time | A<br>Little<br>of the<br>Time | None<br>of the<br>Time |
|---|---|---|---|---|---|---|
| f. Have you felt | 1 | 2 | 3 | 4 | 5 | 6 |
| downhearted and blue? | | | | | | |
| g. Did you feel worn out? | 1 | 2 | 3 | 4 | 5 | 6 |
| h. Have you been a happy | 1 | 2 | 3 | 4 | 5 | 6 |
| person? | | | | | | |
| i. Did you feel tired? | 1 | 2 | 3 | 4 | 5 | 6 |

| 10. During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with your social activities (like visiting with friends, relatives, etc.)? (Circle One Number) | |
|---|---|
| All of the time | 1 |
| Most of the time | 2 |
| Some of the time | 3 |
| A little of the time | 4 |
| None of the time | 5 |

# 11. How TRUE or FALSE is each of the following statements for you.(Circle One Number on Each Line)

| | Definitely | Mostly | Don't | Mostly | Definitely |
|---|---|---|---|---|---|
| | True | True | Know | False | False |
| a. I seem to get sick a little easier than other people | 1 | 2 | 3 | 4 | 5 |
| b. I am as healthy as<br>anybody I know | 1 | 2 | 3 | 4 | 5 |
| c. I expect my health to get worse | 1 | 2 | 3 | 4 | 5 |
| d. My health is excellent | 1 | 2 | 3 | 4 | 5 |

#### **QUICK DEMENTIA RATING SYSTEM (QDRS)**

These next questions are somewhat personal and will help us understand the severity of your symptoms. Please find a private space.

The following descriptions characterize changes in cognitive and functional abilities. Please compare yourself now to how you used to be—the key feature is change. Choose one answer for each category that best fits you. (Note – not all descriptions need to be present to choose an answer.) (for each category there are 5 levels of severity of change)

Which category best describes your:

| | Trinon dategory boot accornace years | |
|---|---|---|
| 1. | Memory and recall | |
| | No obvious memory loss or inconsistent forgetfulness that does not interfere with function in | 0 |
| | everyday activities | |
| | Consistent mild forgetfulness or partial recollection of events that may interfere with performing | 0.5 |
| | everyday activities; repeats questions/statements, misplaces items, forgets appointments | |
| | Mild to moderate memory loss; more noticeable for recent events; interferes with performing everyday activities | 1 |
| | Moderate to severe memory loss; only highly learned information remembered; new information rapidly forgotten | 2 |
| | Severe memory loss, almost impossible to recall new information; long-term memory may be | 3 |
| | affected | |
| 2. | Orientation | |
| | Fully oriented to person, place, and time nearly all the time | 0 |
| | Slight difficulty in keeping track of time; may forget day or date more frequently than in the past | 0.5 |
| | Mild to moderate difficulty in keeping track of time and sequence of events; forgets month or year; oriented to familiar places but gets confused outside familiar areas; gets lost or wanders | 1 |
| | Moderate to severe difficulty, usually disoriented to time and place (familiar and unfamiliar); | 2 |
| | frequently dwells in past Only oriented to their name, although may recognize family members | 3 |
| 3. | | 3 |
| 5. | Solves everyday problems without difficulty; handles personal business and financial matters well; | 0 |
| | decision-making abilities consistent with past performance | |
| | Slight impairment or takes longer to solve problems; trouble with abstract concepts; decisions still sound | 0.5 |
| | Moderate difficulty with handling problems and making decisions; defers many decisions to others; | 1 |
| | social judgment and behavior may be slightly impaired; loss of insight | • |
| | Severely impaired in handling problems, making only simple personal decisions; social judgment and behavior often impaired; lacks insight | 2 |
| | Unable to make decisions or solve problems; others make nearly all decisions for patient | 3 |
| 4. | | |
| | Independent in function at the usual level of performance in profession, shopping, community and | 0 |
| | religious activities, volunteering, or social groups | |
| | Slight impairment in these activities compared with previous performance; slight change in driving skills; still able to handle emergency situations | 0.5 |
| | Unable to function independently but still may attend and be engaged; appears "normal" to others; notable changes in driving skills; concern about ability to handle emergency situations | 1 |
| | No pretense of independent function outside the home; appears well enough to be taken to activities outside the family home but generally needs to be accompanied | 2 |
| | No independent function or activities; appear too ill to be taken to activities outside the home | 3 |

| 5. | Function at home and hobby activities | |
|---|---|---|
| | Chores at home, hobbies and personal interests are well maintained compared with past | 0 |
| | performance | |
| | Slight impairment or less interest in these activities; trouble operating appliances (particularly new | 0.5 |
| | purchases) | |
| | Mild but definite impairment in home and hobby function; more difficult chores or tasks abandoned; | 1 |
| | more complicated hobbies and interests given up | |
| | Only simple chores preserved, very restricted interest in hobbies which are poorly maintained | 2 |
| | No meaningful function in household chores or with prior hobbies | 3 |
| 6. | Toiletting and personal hygiene | |
| | Fully capable of self-care (dressing, grooming, washing, bathing, toileting) | 0 |
| | Slight changes in abilities and attention to these activities | 0.5 |
| | Needs prompting to complete these activities but may still complete independently | 1 |
| | Requires some assistance in dressing, hygiene, keeping of personal items; occasionally incontinent | 2 |
| | Requires significant help with personal care and hygiene; frequent incontinence | 3 |
| 7. | Behavior and personality changes | |
| | Socially appropriate behavior in public and private; no changes in personality | 0 |
| | Questionable or very mild changes in behavior, personality, emotional control, appropriateness of | 0.5 |
| | choices | |
| | Mild changes in behavior or personality | 1 |
| | Moderate behavior or personality changes, affects interactions with others; may be avoided by | 2 |
| | friends, neighbors, or distant relatives | |
| | Severe behavior or personality changes; making interactions with others often unpleasant or | 3 |
| _ | avoided | |
| 8. | Language and communication abilities | |
| | No language difficulty or occasional word searching; reads and writes as in the past | 0 |
| | Consistent mild word finding difficulties, using descriptive terms or takes longer to get point across, | 0.5 |
| | mild problems with comprehension, decreased conversation; may affect reading and writing | 4 |
| | Moderate word finding difficulty in speech, cannot name objects, marked reduction in work | 1 |
| | production; reduced comprehension, conversation, writing, and/or reading | 0 |
| | Moderate to severe impairments in speech production or comprehension; has difficulty in | 2 |
| | communicating thoughts to others; limited ability to read or write | 3 |
| _ | Severe deficits in language and communication; little to no understandable speech is produced | 3 |
| 9. | Mood No changes in mood, interest, or motivation level | 0 |
| | No changes in mood, interest, or motivation level | 0 |
| | Occasional sadness, depression, anxiety, nervousness, or loss of interest/motivation | 0.5 |
| | Daily mild issues with sadness, depression, anxiety, nervousness, or loss of interest/motivation | 2 |
| | Moderate issues with sadness, depression, anxiety, nervousness, or loss of interest/motivation | |
| 40 | Severe issues with sadness, depression, anxiety, nervousness, or loss of interest/motivation Attention and concentration | 3 |
| 10 | | 0 |
| - | Normal attention, concentration, and interaction with his or her environment and surroundings | 0 |
| | Mild problems with attention, concentration, and interaction with environment and surroundings, may | 0.5 |
| | appear drowsy during day Moderate problems with attention and concentration, may have staring spells or spend time with | 1 |
| | | ' |
| | eyes closed, increased daytime sleepiness Significant portion of the day is spend sleeping, not paying attention to environment, when having a | 2 |
| | conversation may say things that are illogical or not consistent with topic | 3 |
| <u></u> | Limited to no ability to pay attention to external environment or surroundings | <u> </u> |

Total QDRS score:

- 2.0 to 6.0 = CDR 0.5 (MCI) -- Eligible
- 6.5 to 12.5 = CDR 1 (mild)-- Eligible
- 13.0 to 17.5 = CDR 2 (moderate)
- ≥18.0 = CDR 3 (severe)

If the QDRS score is 6.5 to 12.5, they are eligible. Otherwise: [1]

## **STOP-BANG Sleep Apnea Questionnaire**

| Name | Height | Weight |
|---|---|---|
| Age Male / Female | | |
| STOP | | |
| Do you SNORE loudly (louder than talking or loud (enough to be heard through closed doors)? | Yes | No |
| Do you often feel TIRED, fatigued, or sleepy during daytime? | Yes | No |
| Has anyone OBSERVED you stop breathing during your sleep? | Yes | No |
| Do you have or are you being treated for high blood PRESSURE? | Yes | No |
| BANG | | |
| BMI more than 35kg/m2? | Yes | No |
| AGE over 50 years old? | Yes | No |
| NECK circumference > 16 inches (40cm)? | Yes | No |
| GENDER: Male? | Yes | No |
| TOTAL SCORE | | |

High risk of OSA: Yes 5-8

Intermediate risk of OSA: Yes 3 - 4

Low risk of OSA: Yes 0 - 2